CLINICAL TRIAL: NCT00241722
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase 3 Study to Evaluate Long-Term Safety and Efficacy of Alvimopan 0.5mg Twice Daily for 12 Months for the Treatment of Opioid-Induced Bowel Dysfunction in Adults Taking Opioid Therapy for Persistent Non-Cancer Pain
Brief Title: Long-Term Safety Evaluation Of Treatment Of Constipation Due To Opioids Being Taken For Persistent Non-Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3753-013; SB-767905/014 (Other: Cubist Study Number)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Bowel Dysfunction; Constipation
Keywords: bowel dysfunction; constipation; gastrointestinal; opioids; pain; non-cancer pain; opioid-induced
MeSH Terms: conditions — Intestinal Diseases; Constipation; Pain | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Alvimopan 0.5 mg Twice Daily (BID) (Experimental): 0.5 milligrams (mg) of alvimopan was administered orally twice daily (BID) for 12 months.
  Interventions: Drug: Alvimopan
- Placebo (Placebo Comparator): Placebo was administered orally BID for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alvimopan
  Arms: Alvimopan 0.5 mg Twice Daily (BID)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Adults who are taking opioid therapy for persistent non-cancer pain and have resulting opioid-induced bowel dysfunction (OBD) will be randomized (1:1) to alvimopan or placebo. The primary objective of this Phase 3 long-term safety study is to compare alvimopan with placebo for safety and tolerability in the treatment of OBD. Participants will be required to attend 8 clinic visits over approximately 1 year.

ELIGIBILITY:
Inclusion criteria:

* Consented to participate in this study.
* Taking opioid therapy for persistent non-cancer pain.
* Has bowel dysfunction mainly due to opioids.
* Has bowel dysfunction since starting opioids as defined by infrequent bowel movements and additional bowel-related symptoms.
* Willing to discontinue laxative therapy (will be provided study-specific standardized laxative if needed).

Exclusion criteria:

* Pregnant, lactating, or planning to become pregnant.
* Not ambulatory.
* Participated in another trial with an investigational drug in the past 30 days.
* Taking opioids for the management of drug addiction or cancer-related pain.
* Severe constipation whereby the subject is at immediate risk of developing serious complications of constipation.
* Gastrointestinal or pelvic disorders known to affect bowel transit, produce gastrointestinal (GI) obstruction, or contribute to bowel dysfunction.
* Human Immunodeficiency Virus (HIV)-infected, has active hepatitis, or has ever been infected with hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2005-08-01 (Actual); Primary Completion 2007-02-01 (Actual); Study Completion 2007-02-01 (Actual)

PRIMARY OUTCOMES:
To compare alvimopan with placebo for long-term safety and tolerability | 12 months

SECONDARY OUTCOMES:
Quality of life, pharmacokinetics, pharmacogenetics (dependent on results from other data) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (200):
- United States (123):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Muscle Shoals, Alabama
  - GSK Investigational Site, Northport, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Pismo Beach, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Stratford, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Chiefland, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Holly Hill, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Dawsonville, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Arlington Heights, Illinois
  - GSK Investigational Site, Bloomington, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Rockford, Illinois
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Pasadena, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Brockton, Massachusetts
  - GSK Investigational Site, Wellesley Hills, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Grand Blanc, Michigan
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Olive Branch, Mississippi
  - GSK Investigational Site, Manchester, Missouri
  - GSK Investigational Site, Nixa, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Dover, New Hampshire
  - GSK Investigational Site, Blackwood, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Concord, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Centerville, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Clinton, Oklahoma
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Oregon City, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Reading, Pennsylvania
  - GSK Investigational Site, Woonsocket, Rhode Island
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Brownwood, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Grand Prairie, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, Lancaster, Texas
  - GSK Investigational Site, Richardson, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Edmonds, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Charleston, West Virginia
- Australia (10):
  - GSK Investigational Site, Broadmeadow, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Carina Heights, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Port Lincoln, South Australia
  - GSK Investigational Site, Toorak Gardens, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
- GSK Investigational Site, Vienna, Austria
- Canada (26):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, North York, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Bonaventure, Quebec
  - GSK Investigational Site, Chandler, Quebec
  - GSK Investigational Site, Drummondville, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- GSK Investigational Site, Ishøj, Denmark
- GSK Investigational Site, Helsinki, Finland
- Hong Kong (4):
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- GSK Investigational Site, Budapest, Hungary
- GSK Investigational Site, Cork, Ireland
- Netherlands (2):
  - GSK Investigational Site, Roosendaal
  - GSK Investigational Site, Utrecht
- New Zealand (3):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Tauranga
- Poland (3):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Wroclaw
- Spain (7):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Ferrol
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Valencia
- Sweden (4):
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Karlstad
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Stockholm
- GSK Investigational Site, Bern, Switzerland
- Taiwan (2):
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- United Kingdom (10):
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Slough, Berkshire
  - GSK Investigational Site, Cardiff, Glamorgan
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Sunbury-on-Thames, Middlesex
  - GSK Investigational Site, Coventry, Warwickshire
  - GSK Investigational Site, Bexhill-on-Sea, East Sussex
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Yaxley, Peterborough